CLINICAL TRIAL: NCT07356323
Title: A Prospective, Single-arm, Trial to Determine Contamination Rates When Using an Antibacterial Incise Drape During Orthopedic Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EM-05-015132
Record Dates: First submitted 2026-01-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty Replacement, Knee; Arthroplasty Total Hip Replacement
Keywords: Chlorohexidine Gluconate; Incise drape; CHG; Ioban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Treatment Arm (Experimental): Subjects undergoing primary hip or knee arthroplasty will have a chlorhexidine gluconate (CHG)-impregnated antimicrobial incise drape applied to the surgical site prior to incision and maintained in place for the duration of the surgical procedure.
  Interventions: Device: 3M™ Ioban™ CHG Chlorhexidine Gluconate Incise Drape (2% w/w CHG)

INTERVENTIONS:
Device: 3M™ Ioban™ CHG Chlorhexidine Gluconate Incise Drape (2% w/w CHG) — A CHG-impregnated antimicrobial incise drape applied to the surgical site prior to incision during primary hip or knee arthroplasty.

SUMMARY:
The goal of this clinical study is to generate data on the intended use of a chlorhexidine gluconate (CHG)-impregnated antimicrobial incise drape. The study includes subjects undergoing primary hip or knee arthroplasty procedures.

The study evaluates the intraoperative performance and safety of the incise drape during surgery, including assessment of contamination and operative characteristics.

Participants will have a CHG-impregnated antimicrobial incise drape applied during their surgical procedure. During surgery, samples will be collected from the operative site to assess potential bacterial contamination.

DETAILED DESCRIPTION:
This is a prospective, single-arm clinical study conducted in the United States in subjects undergoing primary hip or knee arthroplasty. The study evaluates the intraoperative performance and safety of a chlorhexidine gluconate (CHG)-impregnated antimicrobial incise drape used during lower extremity orthopedic surgery.

Safety and intraoperative performance outcomes will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 22 years of age on the day of surgery.
* Subject is scheduled to undergo a unilateral primary arthroplasty procedure on a hip or knee.
* Subject is capable of providing informed consent.
* Subject is willing and able to return for all visits.

Exclusion Criteria:

* Subject is pregnant or lactating prior to surgery.*

  *Women who have had surgical sterilization by a medically accepted method (e.g., tubal ligation, hysterectomy, or oophorectomy) or are post-menopausal, defined as not having menstruation for > 12 months will not be required to undergo pregnancy testing
* Subject is scheduled to undergo a lower extremity bilateral arthroplasty procedure.
* Subject had a previous open knee surgery on the study knee or is scheduled to undergo a revision knee arthroplasty.
* Subject has had a previous surgery for revision femoral acetabular osteotomy or total hip arthroplasty on the study hip.
* Subject is scheduled for lower extremity arthroplasty due to trauma.
* Subject was previously diagnosed with septic arthritis or has a history of infection in the joint.
* Subject has taken any antibiotics within 4 weeks before surgery.
* Subject has an allergy or sensitivity to components of the device (e.g., chlorhexidine gluconate or acrylate-based adhesive).
* Subject is currently enrolled in another trial.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the presence of contamination at the surgical site during the operative procedure. | During surgery
  Assessment of contamination at the surgical site during the operative procedure.

OTHER OUTCOMES:
Percentage of Subjects With Loss of Incise Drape Adherence Greater Than 10 mm During Surgery | During surgery
  The percentage of subjects who experience loss of adherence of the incise drape of more than 10 millimeters (mm) at the incision site during the surgical procedure.
Operative Time | During surgery
  Operative time measured in minutes

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University Health (IU Health), Fishers, Indiana
  - University of Utah Health - Department of Orthopedics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No